CLINICAL TRIAL: NCT02026024
Title: Clinical and Genetic Variations Study of Incretin Based Therapy for Poorly Controlled Type 2 Diabetic Patients
Brief Title: Incretin Based Therapy for Poorly Controlled Type 2 Diabetic Patients
Acronym: IBCT2
Status: Completed | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 102-3596B
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — DNA for sequencing
Oversight: Data Monitoring Committee: No

SUMMARY:
Type 2 diabetes patients have been proved to have decreased of glucagon-like peptide-1 (GLP-1) levels. Incretin based therapy is associated with improved glycemic control by boosting GLP-1 levels . Nevertheless, the clinical effects are in great diversity for poorly controlled Type 2 diabetes patients. This study is designed to understand the pharmacological effects and genetic variation of incretin based therapy on type 2 diabetes.

DETAILED DESCRIPTION:
Background:

Since GLP-1 receptor is encoded by GLP1R ( glucagon-like peptide-1 receptor) gene, individuals may veritably respond to incretion based treatment, depending on the presence or absence of minor alleles characterized by single nucleotide polymorphisms. The genotyping of patients will be performed to compare the genetic factors and the pharmacological effects.

Expected Results: How to select a anti-diabetic drug tailored to the individual becomes more and more important because the enormously increasing classes of treatment modality. This study could be of great help in recommending the best possible agent for an individual, improving the possibility of treatment success, and justifying if the need of expensive drugs in a given patient.

ELIGIBILITY:
Inclusion Criteria:

* i) Age > 20 years old ii)DM (diabetes mellitus) diagnosed > 2 years iii)HbA1c level of 8% to 12% iv) Receiving incretin based therapy at least one month (including either GLP-1 agonist or DPP(dipeptidyl peptidase)-IV inhibitor

Exclusion Criteria:

* Type 1 Diabetes Mellitus

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Poorly Controlled Type 2 Diabetic Patients
Sampling Method: Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
mean amplitude of glycaemic excursions (MAGE) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: CHIA-HUNG LIN, M.D., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan, Taiwan